CLINICAL TRIAL: NCT01866423
Title: Phase 2 Trial of TAK-700 (Also Known as Orteronel) Without Prednisone for Metastatic Castration-Resistant Prostate Cancer
Brief Title: Orteronel in Treating Patients With Metastatic Hormone-Resistant Prostate Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Not progressing toward scientific goals
Sponsor: University of Southern California (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Millennium Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 4P-13-1; NCI-2013-01013 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); IISR-2012-M000668; P30CA014089 (NIH)
Record Dates: First submitted 2013-05-28; First posted 2013-05-31 (Estimated); Results first posted 2017-08-31 (Actual); Last update posted 2017-08-31 (Actual); Status verified 2017-06

CONDITIONS: Adenocarcinoma of the Prostate; Hormone-resistant Prostate Cancer; Recurrent Prostate Cancer; Stage IV Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — orteronel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (orteronel) (Experimental): Patients receive orteronel 300 mg PO BID on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: orteronel; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: orteronel — Given PO
  Other Names: TAK-700
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This phase II trial studies how well orteronel works in treating patients with metastatic hormone-resistant prostate cancer. Orteronel may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess the relationship between circulating tumor cell (CTC)-based androgen receptor (AR) expression level and >=-50% prostate-specific antigen (PSA) decline following 12 weeks of therapy with TAK-700 (orteronel).

SECONDARY OBJECTIVES:

I. To assess changes in PSA and CTC levels and time to PSA progression (best response, decline at 12 weeks as continuous variable, etc.) with or without prior docetaxel-based treatment.

II. To assess measurable disease response and time to radiographic disease progression for castration-resistant prostate cancer (CRPC) with or without prior docetaxel-based treatment.

III. To explore relationships between endocrine and clinical responses.

IV. To confirm the safety of TAK-700 administered without prednisone in patients with metastatic CRPC.

OUTLINE: Patients receive orteronel orally (PO) twice daily (BID) on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed adenocarcinoma of the prostate
* Voluntary written informed consent before performance of any study-related procedure not part of normal medical care, with the understanding that consent may be withdrawn by the subject at any time without prejudice to future medical care
* Patients, even if surgically sterilized (i.e., status post vasectomy), who agree to practice effective barrier contraception during the entire study treatment period and for 4 months after the last dose of study drug, or
* Agree to completely abstain from intercourse
* Serum alanine aminotransferase (ALT) and aspartate aminotransferase (AST) must be =< 2.5 x the upper limit of normal (ULN)
* Total bilirubin =< 1.5 x ULN
* Estimated creatinine clearance using the Cockcroft-Gault formula must be > 40 mL/minute
* Absolute neutrophil count (ANC) >= 1500 cells/microliter
* Platelet count >= 100,000 cells/microliter
* Testosterone < 50 ng/dL
* Screening calculated ejection fraction of >= 50% by multiple gated acquisition (MUGA) scan or echocardiogram; metastatic progression on primary androgen-deprivation therapy (medical or surgical castration)
* Progression requiring a change in oncologic therapy defined by any of the following:

  * Radiographic progression: appearance or increase in measurable lesions on cross-sectional imaging or appearance of one or more new lesions on bone scan * Rising PSA (>= 2 ng/ml) which has risen on two occasions >= 1 week apart
  * Clinical progression evidenced by increased pain or other cancer-related symptoms
* Patients should have recovered from prior oncologic therapies to a Common Terminology Criteria (CTC) grade =< 1 except stable neuropathy or alopecia at National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) grade =< 2; if rapid clinical progression is documented by imaging, changes in PSA, or symptoms, then study treatment can begin >= 2 weeks from prior therapy; otherwise, the following time periods between prior anti-cancer therapies and study treatment day 1 will apply:

  * >= 3 weeks for prior cytotoxic therapies
  * >= 4 weeks for flutamide or nilutamide
  * >= 6 weeks for bicalutamide
  * >= 6 weeks since bone targeted radiopharmaceutical (e.g. samarium-153, radium-223)
* Gonadotropin-releasing hormone (GnRH) agonists (leuprolide acetate, goserelin, etc.) or antagonists (degarelix, etc.) should be continued in patients without surgically-induced castrate androgen levels
* For chemotherapy naïve castration-resistant prostate cancer who are moderately symptomatic or who have hepatic metastasis: subjects must not be a candidate for docetaxel-based chemotherapy.

Exclusion Criteria:

* History of myocardial infarction, unstable symptomatic ischemic heart disease, ongoing arrhythmias of grade > 2 (NCI CTCAE, version 4), thromboembolic events (e.g., deep vein thrombosis, pulmonary embolism, or symptomatic cerebrovascular events), or any other cardiac condition (e.g. pericardial effusion, restrictive cardiomyopathy) within 6 months prior to first dose of study drug; chronic stable atrial fibrillation on stable anticoagulant therapy is allowed
* New York Heart Association class III or IV heart failure
* Electrocardiogram (ECG) abnormalities of:

  * Q-wave infarction, unless identified 6 or more months prior to screening
  * Corrected QT (QTc) interval > 460 msec
* Patient has received other investigational drugs within 28 days before enrollment
* Diagnosed or treated for another malignancy within 2 years of enrollment, with the exception of complete resection of basal cell carcinoma or squamous cell carcinoma of the skin, an in situ malignancy
* Known hypersensitivity to compounds related to TAK-700 or to TAK-700 excipients
* Uncontrolled hypertension despite appropriate medical therapy (blood pressure [BP] of greater than 160 mmHg systolic and 90 mmHg diastolic at 2 separate measurements no more than 60 minutes apart during the screening visit); Note: patients may be rescreened after adjustment of antihypertensive medications
* Known active chronic hepatitis B or C, life-threatening illness unrelated to cancer, or any serious medical or psychiatric illness that could, in the investigator's opinion, potentially interfere with participation in this study
* Likely inability to comply with the protocol or cooperate fully with the investigator and site personnel
* Known gastrointestinal (GI) disease or GI procedure that could interfere with the GI absorption or tolerance of TAK-700, including difficulty swallowing tablets
* Prior treatment with >= 3 lines of cytotoxic chemotherapy for metastatic prostate cancer
* Prior treatment with TAK-700

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2013-10-25 (Actual); Primary Completion 2015-07-23 (Actual); Study Completion 2016-07-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mitchell Gross, Principal Investigator — University of Southern California
Locations (1):
- USC Norris Comprehensive Cancer Center, Los Angeles, California, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited at the University of Southern California (USC) medical clinics from December 2013 to February 2014. Due to results of two phase III clinical trials in metastatic, castration resistant prostate cancer (mCRPC), the sponsor determined that the drug has not demonstrated a clinical profile sufficient to move forward in mCRPC.
Pre-assignment Details: The trial had no pre-assignment criteria. All subjects were given the same treatment.
Groups:
- Treatment (Orteronel): Patients receive orteronel 300 mg PO BID (twice a day) on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  orteronel: Given PO
  laboratory biomarker analysis: Correlative studies
Period: Overall Study
Arm/Group | Treatment (Orteronel)
Started | 4
Completed | 0
Not Completed | 4
Not completed — Lack of Efficacy | 3
Not completed — Sponsor Decision | 1

BASELINE CHARACTERISTICS:
Groups:
- Treatment (Orteronel): Patients receive orteronel 300 mg PO twice daily (BID) on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  orteronel: Given PO
  laboratory biomarker analysis: Correlative studies
Arm/Group | Treatment (Orteronel)
Number analyzed (Participants) | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 4
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 4

OUTCOME MEASURES:

1. Primary Outcome: Androgen Receptor (AR) Protein Expression Levels in CTCs
Description: The two-sample t-test will be used. Once association between AR protein expression levels and response is established, graphical methods such as receiver-operator curves (ROC) or more quantitative methods such as the maximal chi-square method to determine whether there might be a cut-point with either great sensitivity or great specificity (or both) for identifying a cohort with either a high or low likelihood of prostate-specific antigen (PSA) response.
Time Frame: Up to 4 weeks
Population: Only 4 patients were accrued to this trial. No data analysis was performed.
Arm/Group | Treatment (Orteronel)
Number analyzed (Participants) | 0

2. Primary Outcome: PSA Response, Defined as Occurrence of PSA Decline to Greater Than or Equal to 50% From Baseline
Description: Standard descriptive methods will be used to summarize PSA. Values will be tabulated as outlined in the Prostate Cancer Working Group 2 (PCWG2) criteria and presented as Kaplan-Meier survival curves, as appropriate.
Time Frame: At 12 weeks
Population: Only 4 patients were accrued to this trial. No data analysis was performed.
Arm/Group | Treatment (Orteronel)
Number analyzed (Participants) | 0

3. Secondary Outcome: Best PSA Response
Description: Values will be tabulated as outlined in the PCWG2 criteria and presented as Kaplan-Meier survival curves, as appropriate.
Time Frame: Up to 24 weeks
Population: Only 4 patients was accrued to this trial. No data analysis was performed.
Arm/Group | Treatment (Orteronel)
Number analyzed (Participants) | 0

4. Secondary Outcome: Absolute Change in PSA
Description: as for outcome 3
Time Frame: Baseline to 24 weeks
Population: Only 4 patients was accrued to this trial. No data analysis was performed.
Arm/Group | Treatment (Orteronel)
Number analyzed (Participants) | 0

5. Secondary Outcome: Overall Response Rate Using Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1 and PCWG2 Criteria
Description: Response will be tabulated descriptively with 95% confidence intervals (CIs) and Kaplan-Meier survival curves, as appropriate.
Time Frame: Up to 3 years
Population: Only 4 patients was accrued to this trial. No data analysis was performed.
Arm/Group | Treatment (Orteronel)
Number analyzed (Participants) | 0

6. Secondary Outcome: Duration of Response Using RECIST Version 1.1 and PCWG2 Criteria
Description: Response will be tabulated descriptively with 95% CIs and Kaplan-Meier survival curves, as appropriate.
Time Frame: Up to 3 years
Population: Only 4 patients was accrued to this trial. No data analysis was performed.
Arm/Group | Treatment (Orteronel)
Number analyzed (Participants) | 0

7. Secondary Outcome: Number of Participants With Grade 3 or Higher Toxicity
Description: Summary of grade 3 (per Common Terminology Criteria for Adverse Events (CTCAE v4.0) or higher toxicities which generally is described as a severe reaction or symptom.
Time Frame: 30 days
Population: Tracked during treatment period until 30 days after last dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Orteronel)
Number analyzed (Participants) | 4
Participants | 1

ADVERSE EVENTS:
Time Frame: Days 1, 8, 15, 21 of each cycle and treatment end (30 days after last dose or start of new treatment).
Arm/Group | Treatment (Orteronel)
All-Cause Mortality (participants affected / at risk) | 0/4
Serious Adverse Events (participants affected / at risk) | 1/4
Other Adverse Events (participants affected / at risk) | 3/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Orteronel) (N=4)
Abdominal Pain (Gastrointestinal disorders) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 1 (1)
Hypertension (Vascular disorders) | 1 (1)
Platelet count decreased (Investigations) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Orteronel) (N=4)
Abodminal Pain (Gastrointestinal disorders) | 2 (2)
Anorexia (Metabolism and nutrition disorders) | 3 (3)
Activated partial thromboplastin time prolonged (Investigations) | 1 (1)
Adrenal insufficiency (Endocrine disorders) | 1 (1)
Alkaline phosphatase increased (Investigations) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 1 (2)
Aspartate Aminotransferase increased (Investigations) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (2)
Bruising (Injury, poisoning and procedural complications) | 1 (1)
Chest pain - cardiac (Cardiac disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 2 (4)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (4)
Creatinine increased (Investigations) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (2)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Electrocardiogram QT corrected interval prolonged (Investigations) | 1 (1)
Fatigue (General disorders) | 3 (4)
Fever (General disorders) | 2 (2)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
Hematuria (Renal and urinary disorders) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 2 (2)
Hyperkalemia (Metabolism and nutrition disorders) | 1 (1)
Hypertension (Vascular disorders) | 1 (1)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (2)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1)
Hypophosphatemia (Metabolism and nutrition disorders) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1)
Libido decreased (Psychiatric disorders) | 2 (3)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 3 (3)
Neutrophil count decreased (Investigations) | 1 (1)
Pain (General disorders) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (2)
Platelet count decreased (Investigations) | 1 (2)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Stomach pain (Gastrointestinal disorders) | 2 (2)
Tooth infection (Infections and infestations) | 1 (1)
Toothache (Gastrointestinal disorders) | 1 (1)
Urinary frequency (Renal and urinary disorders) | 1 (2)
Vomiting (Gastrointestinal disorders) | 2 (2)
White blood cell decreased (Investigations) | 1 (1)

LIMITATIONS AND CAVEATS:
The trial was terminated early due to the discontinuation of the development program for the study drug, TAK-700 (orteronel) for prostate cancer.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes